CLINICAL TRIAL: NCT04844606
Title: A Master Protocol for a Phase 3, Multicenter, Open-label, Long-term Extension Study to Evaluate the Long-term Efficacy and Safety of Mirikizumab in Children and Adolescents With Moderate-to-severe Ulcerative Colitis or Crohn's Disease
Brief Title: A Master Protocol (AMAZ): A Study of Mirikizumab (LY3074828) in Pediatric Participants With Ulcerative Colitis or Crohn's Disease (SHINE-ON)
Acronym: SHINE-ON
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16633; I6T-MC-AMAZ (Other: Eli Lilly and Company); 2020-005311-49 (EudraCT Number); ISA-1 UC (Other: Eli Lilly and Company); ISA-2 CD (Other: Eli Lilly and Company); ISA-3 UC (Other: Eli Lilly and Company); ISA-4 CD (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-04-12; First posted 2021-04-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis; Ulcerative Colitis Chronic; Inflammatory Bowel Diseases; Crohn's Disease
Keywords: Pediatric Ulcerative Colitis; Pediatric Crohn's Disease; Pediatric UC; Pediatric CD
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases; Crohn Disease; Pediatric ulcerative colitis; Pediatric Crohn's disease | interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Mirikizumab Dose 1 for UC (Experimental): Dose 1 of Mirikizumab is administered subcutaneously (SC)
  Dosing is based on the participant's weight.
  Interventions: Drug: Mirikizumab
- Mirikizumab Dose 2 for UC (Experimental): Dose 2 of Mirikizumab is administered SC
  Dosing is based on the participant's weight.
  Interventions: Drug: Mirikizumab
- Mirikizumab Dose 3 for UC (Experimental): Dose 3 of Mirikizumab is administered SC
  Dosing is based on the participant's weight.
  Interventions: Drug: Mirikizumab
- Mirikizumab Dose 4 for CD (Experimental): Dose 4 of Mirikizumab is administered SC
  Dosing is based on the participant's weight.
  Interventions: Drug: Mirikizumab
- Mirikizumab Dose 5 for CD (Experimental): Dose 5 of Mirikizumab is administered SC
  Dosing is based on the participant's weight.
  Interventions: Drug: Mirikizumab
- Mirikizumab Dose 6 for CD (Experimental): Dose 6 of Mirikizumab is administered SC
  Dosing is based on the participant's weight.
  Interventions: Drug: Mirikizumab
- Mirikizumab Dose 7 for UC or CD (Experimental): Intravenous (IV) rescue dosing, if response is lost.
  Interventions: Drug: Mirikizumab

INTERVENTIONS:
Drug: Mirikizumab — Administered SC
  Other Names: LY3074828
  Arms: Mirikizumab Dose 1 for UC; Mirikizumab Dose 2 for UC; Mirikizumab Dose 3 for UC; Mirikizumab Dose 4 for CD; Mirikizumab Dose 5 for CD; Mirikizumab Dose 6 for CD
Drug: Mirikizumab — Administered IV
  Other Names: LY3074828
  Arms: Mirikizumab Dose 7 for UC or CD

SUMMARY:
The main purpose of this study is to evaluate the long-term efficacy of mirikizumab in pediatric participants with ulcerative colitis (UC) or Crohn's disease (CD). The study will last about 172 weeks and may include up to 44 visits. Additional treatment may be available to participants via a Continued Access Period.

ELIGIBILITY:
Inclusion Criteria:

* Participants from originating studies (I6T-MC-AMBA [NCT05784246], I6T-MC-AMBU [NCT04004611], I6T-MC-AMAM [NCT03926130]) , I6T-MC-AMAY [NCT05509777]) who would, in the opinion of the investigator, derive clinical benefit from further treatment with mirikizumab
* Participants from prior studies who have completed assessments and procedures at last visit of originating study and remain on study drug treatment.
* Female participants must agree to contraception requirements.

Exclusion Criteria:

* Participants must not have developed a serious adverse event (SAE) or Adverse Event (AE) in originating study or developed other condition before first visit of Study AMAZ that continued treatment with mirikizumab would present an unreasonable risk for the participant.
* Participants must not have had permanently or temporarily stopped study drug in the originating study, such that restarting mirikizumab would pose an unacceptable risk for the participant in Study AMAZ.
* Participants must not have an unstable or uncontrolled illness that would potentially affect participant safety.
* Participants must not be enrolled in the study if, for any reason, being in the study would compromise the participant's safety or confound data interpretation.
* Participants must not have adenomatous polyps that have not been removed.
* Participants must not be pregnant or breastfeeding.

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with UC in Modified Mayo Score (MMS) Clinical Remission | Week 52
  Clinical Remission based on the MMS
Percentage of Participants with CD in Pediatric Crohn's Disease Activity Index (PCDAI) Clinical Remission | Week 52
  Clinical Remission based on the PCDAI

SECONDARY OUTCOMES:
Percentage of Participants with UC in MMS Clinical Response | Week 52
  Clinical Response based on the MMS
Percentage of Participants with CD in PCDAI Clinical Response | Week 52
  Clinical Response based on the PCDAI
Percentage of Participants with UC in Pediatric Ulcerative Colitis Activity Index (PUCAI) Clinical Response | Week 52
  Clinical Response based on the PUCAI
Percentage of Participants with UC in PUCAI Clinical Remission | Week 52
  Clinical Response based on the PUCAI
Percentage of Participants with UC in Endoscopic Remission | Week 52
  Endoscopic Remission based on the Endoscopic Subscore (ES)
Percentage of Participants with CD in Endoscopic Remission | Week 52
  Endoscopic Remission in Participants based on the Simple Endoscopic Score for Crohn's Disease (SES-CD)
Percentage of Participants with UC in Endoscopic Response | Week 52
  Endoscopic Response in Participants based on the ES
Percentage of Participants with CD in Endoscopic Response | Week 52
  Endoscopic Response based on the SES-CD
Percentage of Participants with UC in having Endoscopic Subscore = 0 | Week 52
  Endoscopic Remission when ES = 0
Percentage of Participants with UC Histologic-Endoscopic Mucosal Remission | Week 52
  Histologic remission based on histology scoring and endoscopic remission based on endoscopy score
Percentage of Participants with CD Achieving Histologic Remission | Week 52
  Histologic remission based on histology scoring
Percentage of Participants with UC in Corticosteroid-free Remission Without Surgery | Week 52
  Corticosteroid-free Remission based on MMS in participants who did not have an ulcerative colitis (UC)-related surgery
Percentage of Participants with CD in Corticosteroid-free Remission Without Surgery | Week 52
  Corticosteroid-free Remission based on PCDAI in participants who did not have Crohn's disease (CD-related surgery)
Time to First Dose of Corticosteroid Among Participants with UC Entering Study AMAZ Not on Corticosteroids | Week 0 to Week 52
Percentage of Participants Who Achieve both Clinical Remission by PCDAI and Endoscopic Response | Week 52
Change from Baseline Over Time in C-reactive Protein, High Sensitivity (hsCRP) | Baseline, Week 0 to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (61):
- United States (10):
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Emory University School of Medicine, Atlanta, Georgia
  - Children's Center for Digestive Health Care, LLC, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Waltham, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cook Children's Medical Center, Fort Worth, Texas
  - Pediatric Specialists of Virginia, Fairfax, Virginia
- Medizinische Universität Wien, Vienna, Austria
- Belgium (5):
  - UZ Brussel, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Antwerp University Hospital, Edegem
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Brazil (7):
  - Centro de Pesquisa Sao Lucas, Campinas
  - Hospital Pequeno Príncipe / Associação Hospitalar de Proteção à Infância, Curitiba
  - Universidade Federal de Goias, Goiânia
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Hospital Universitario Cassiano Antonio de Moraes, Vitória
  - Integral Pesquisa e Ensino, Votuporanga
- The Hospital for Sick Children, Toronto, Canada
- Germany (2):
  - Universitätsmedizin Johannes Gutenberg Universität Mainz, Mainz
  - Dr. von Haunersches Kinderspital, Munich
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
  - Yitzhak Shamir Medical Center, Ẕerifin
- Italy (6):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - Ospedale Maggiore Azienda USL di Bologna, Bologna
  - Azienda Ospedaliera Universitaria Meyer IRCCS, Florence
  - Ospedale dei Bambini Vittore Buzzi, Milan
  - AOU Policlinico Umberto I, Roma
  - Ospedale Pediatrico Bambino Gesù IRCCS, Rome
- Japan (4):
  - Institute of Science Tokyo Hospital, Bunkyō
  - Juntendo University Hospital, Bunkyō City
  - Tsujinaka Hospital - Kashiwanoha, Kashiwa
  - Yokohama City University Medical Center, Yokohama
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- Norway (2):
  - Akershus Universitetssykehus, Lørenskog
  - St. Olavs Hospital, Trondheim
- Poland (5):
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Twoja Przychodnia SCM, Szczecin
  - Medical Network Spółka z o.o. WIP Warsaw IBD Point Profesor Kierkuś, Warsaw
  - Centrum Zdrowia Dziecka w Warszawie, Warsaw
  - Centrum Medyczne Oporów, Wroclaw
- Portugal (2):
  - 2Ca Braga, Braga
  - Centro Hospitalar de Sao Joao - Hospital de Sao Joao, Porto
- South Korea (3):
  - Kyungpook National University Chilgok Hospital, Deagu
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
  - Hospital Universitari Parc Tauli, Sabadell
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (3):
  - Royal London Hospital, London
  - The John Radcliffe Hospital, Oxford
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Master Protocol (AMAZ): A Study of Mirikizumab (LY3074828) in Pediatric Participants With Ulcerative Colitis or Crohn's Disease (SHINE-ON) — https://trials.lillytrialguide.com/en-US/trial/6Fqthjwf4KUkJi8EyTQv5A